CLINICAL TRIAL: NCT05858411
Title: Evaluation of the Efficacy of rhPDGF as an Adjunct to Non-surgical Periodontal Therapy of Intrabony Defects: a Randomized Controlled Clinical Trial
Brief Title: Efficacy of rhPDGF as an Adjunct to Non-surgical Periodontal Therapy of Intrabony Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Full time professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21042023
Record Dates: First submitted 2023-04-21; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Periodontal Diseases; Periodontal Attachment Loss; Pocket, Periodontal; Intrabony Periodontal Defect
Keywords: rhPDGF; Growth factors; Periodontal regeneration
MeSH Terms: conditions — Periodontal Diseases; Periodontal Attachment Loss; Periodontal Pocket

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SRP+rhPDGF (Experimental): After SRP the infrabony defect will be filled with a collagen sponge soaked in rhPDGF.
  Interventions: Procedure: SRP+rhPDGF
- SRP+ collagen sponge (Active Comparator): After SRP the infrabony defect will be filled with a collagen sponge soaked in saline solution.
  Interventions: Procedure: SRP+collagen sponge
- SRP alone (Active Comparator): SRP alone will be performed.
  Interventions: Procedure: SRP alone

INTERVENTIONS:
Procedure: SRP+rhPDGF — The infrabony defect will be debrided with the use of fine ultrasonic tips and mini hand instruments and will be treated with the application of a collagen sponge soaked in rhPDGF.
  Arms: SRP+rhPDGF
Procedure: SRP+collagen sponge — The infrabony defect will only be debrided with the use of fine ultrasound tips and mini hand instruments and will be treated with the application of a collagen sponge soaked in saline solution.
  Arms: SRP+ collagen sponge
Procedure: SRP alone — The infrabony defect will only be debrided with the use of fine ultrasound tips and mini hand instruments and no further treatment will be performed.
  Arms: SRP alone

SUMMARY:
The aim of the present study is to clinically and radiographically evaluate the efficacy of recombinant human platelet-derived growth factor (rhPDGF) in intrabony defects following scaling and root planing (SRP).

This study will be designed as a randomized clinical trial of 12-month duration. A total of 51 patients (each with a single infrabony defect) will be recruited and randomly equally distributed into 3 groups: an experimental group treated with SRP and rhPDGF, a first control group treated with SRP and collagen sponge and a second control group treated with SRP alone.

Each defect will be treated with an ultrasonic scaler with dedicated thin tips for supra- and subgingival debridement associated with hand instrumentation under local anesthesia. Caution will be taken to preserve the stability of soft tissues. Following SRP, experimental and control sites will be randomly chosen. The test sites will be treated by inserting a collagen plug soaked for at least 15 minutes in a 1.5cc solution containing hPDGF-BB. In the first control group the infrabony defects will be treated with SRP and a collagen sponge soaked in saline solution. In the second control sites no further treatment will be carried out.

Pre- and post-treatment clinical measurements were performed by an examiner blinded to the treatment modalities using a graded periodontal probe (HuFriedy UNC 15). Before the treatment and at 6 and 12 months post-treatment, all patients were examined by measuring the clinical attachment level, probing depth, gingival recession, full-mouth plaque score and bleeding on probing.

Standardized radiographs of selected study sites will be taken at baseline and at the 6 and 12 months follow-up visits using the long-cone technique with a customized holder and a thermoplastic occlusal reference to allow reproducible positioning. All radiographs will be analysed by a dedicated dental software (Carestream Dental LLC Atlanta, GA, USA) to make linear measurements. The defect bone level (DBL), the defect angle (DA) and the radiographic defect area (RDA) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of periodontitis stage III or IV (grades A to C),
* non-smokers or former smokers who quit at least 1 year ago, and
* had not received any periodontal treatment in the 3 months prior to recruitment;
* Presence of at least 1 Infrabony defect (PPD ≥ 5 mm with infrabony defect depth of ≥3mm at screening radiograph);
* One and two wall infrabony defects at screening radiograph and periodontal charting.
* Signed informed consent.

Exclusion Criteria:

* Presence of uncontrolled systemic diseases that could affect treatment outcomes such as diabetes mellitus with an HbA1C>7%, rheumatoid arthritis or any form of immunosuppression;
* Subjects requiring antibiotic prophylaxis;
* 3-wall infrabony defects;
* Patients that had received systemic or local delivery of antibiotic therapy 6 weeks before enrollment;
* Presence of furcation defect;
* Chronic intake of NSAIDs or steroids, currently;
* Patients undergoing orthodontic treatment, having removable prosthetic appliances, pregnancy, tumors of the oral cavity or the presence of any psychiatric condition that could affect participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-05-08 (Estimated); Primary Completion 2024-12-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Defect Bone Level (DBL) | 12 months
  Distance between the cemento-enamel junction (CEJ) and the bottom of the defect (BD)
Clinical Attachment Level (CAL) | 12 months
  Distance between the CEJ and the bottom of the pocket

SECONDARY OUTCOMES:
Pocket Probing Depth (PPD) | 12 months
  Distance between the gingival margin and the bottom of the pocket.
Gingival Recession (GR) | 12 months
  Distance between the CEJ and the gingival margin.
Defect Angle (DA) | 12 months
  Angle between the long axis of the tooth and the interproximal wall of the infrabony defect.
Radiographic Defect Area | 12 months
  Area of the triangle defined by: side passing through the top of the interproximal ridge and perpendicular to the long axis of the tooth, side passing through the bottom of the defect and the intersection of the previous side with the root of the tooth, side passing through the top of the ridge and the bottom of the defect.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Paolantonio, DDS, MD, Study Chair — University 'G. D'Annunzio' of Chieti

IPD SHARING:
Plan to Share IPD: No